CLINICAL TRIAL: NCT02084953
Title: A Randomized, Double-Blinded, Positive-Controlled, Placebo-Controlled, 3-Way Crossover Study to Determine the Electrocardiographic Effects of BMS-791325 in Healthy Subjects
Brief Title: Study to Determine the Effect of BMS-791325 on the ECG QTcF Interval in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: AI443-112
Record Dates: First submitted 2014-03-10; First posted 2014-03-12 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ARM A: BMS-791325 (Experimental): BMS-791325 600 mg tablet orally on 1st and 2nd day, then 900 mg on the 3rd day once a day for 3 days
  Interventions: Drug: BMS-791325
- ARM B: Moxifloxacin (Active Comparator): Moxifloxacin 400mg tablet orally once on third day
  Interventions: Drug: Moxifloxacin
- ARM C: Placebo matching BMS-791325 (Placebo Comparator): Placebo matching BMS-791325 0 mg tablet orally once daily for 3 days
  Interventions: Drug: Placebo matching BMS-791325

INTERVENTIONS:
Drug: BMS-791325
  Arms: ARM A: BMS-791325
Drug: Moxifloxacin
  Other Names: Avelox®
  Arms: ARM B: Moxifloxacin
Drug: Placebo matching BMS-791325
  Arms: ARM C: Placebo matching BMS-791325

SUMMARY:
The purpose of this study is to determine whether BMS-791325 has an effect on the electrocardiogram (ECG) interval QT corrected for Fridericia's method (QTcF).

DETAILED DESCRIPTION:
Primary Purpose: Other: This Phase 1 study is a clinical pharmacology thorough QT study.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Healthy men and women, ages 18 to 49 yr old
* BMI 18 to 32
* Women must not be pregnant or breastfeeding

Exclusion Criteria:

* Any significant acute or chronic medical illness
* A personal history of clinically relevant cardiac disease, symptomatic or asymptomatic arrhythmias, presyncope or syncopal episodes, or additional risk factors for torsades de pointes (eg, heart failure)
* History of hypokalemia, personal history or family history of prolonged QT interval, or family history of sudden cardiac death at a young age
* History of biliary disorders, including Gilbert's disease or Dubin-Johnson disease
* Inability to swallow multiple tablets consecutively
* Any of the following on 12-lead electrocardiogram (ECG) prior to study drug administration: PR ≥ 210 msec, QRS ≥ 120 msec, QT ≥ 500 msec, QTcF ≥ 450 msec, Heart Rate (HR) < 45 bpm
* Second or third degree heart block prior to study drug
* Positive urine screen for drugs of abuse
* Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, or Human Immunodeficiency Virus (HIV)-1, -2 antibody
* Any of the following lab results outside of the ranges specified below prior to dosing: Alanine aminotransferase (ALT) > upper limit of normal (ULN), Aspartate aminotransferase (AST) > ULN, Total bilirubin > ULN, Direct bilirubin > ULN, Creatinine > ULN, Serum potassium < lower limit of normal (LLN), Serum magnesium < LLN
* History of allergy to Moxifloxacin, BMS-791325, nonstructural protein 5B (NS5B) non-nucleoside inhibitors or related compounds

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Difference from placebo of BMS-791325 in time-matched change from baseline (Day -1 on the study) to Day 3 of each period (ΔΔQTcF) at postdose extraction times for the QTcF | Approximately 28 days

SECONDARY OUTCOMES:
ΔΔHR, ΔΔPR, ΔΔQRS, ΔΔQT | Approximately 28 days
  Difference from placebo in time-matched change from baseline (Day -1) to Day 3 at postdose extraction times in the ECG-derived RR or HR and other ECG intervals (PR, QRS, QT). QT is the unadjusted QT interval
Number and percent of subjects having a within-period maximum HR, PR, QRS, QT, QTcF, ΔQT and ΔQTcF within prespecified categories | Approximately 28 days
Relationship between plasma concentrations of BMS-791325, BMS-794712, and BMS-948158, and the corresponding ΔΔQTcF | Approximately 28 days
Maximum observed concentration (Cmax) of BMS-791325, BMS-794712, and BMS-948158 | 43 timepoints up to day 26
Time of maximum observed concentration (Tmax) of BMS-791325, BMS-794712, and BMS-948158 | 43 timepoints up to day 26
Area under the concentration-time curve in one dosing interval (AUC(TAU)) of BMS-791325, BMS-794712, and BMS-948158 | 43 timepoints up to day 26
Apparent total oral clearance (CLT/F) of BMS-791325, BMS-794712, and BMS-948158 | 43 timepoints up to day 26
Terminal phase plasma half life (T-HALF) of BMS-791325, BMS-794712, and BMS-948158 | 43 timepoints up to day 26
AUC(TAU) metabolic ratios of BMS-791325, BMS-794712, and BMS-948158 | 43 timepoints up to day 26
Incidence of AEs, SAEs, AEs leading to discontinuation and death, marked laboratory abnormalities, findings on 12-lead safety ECG measurements and physical examination, and abnormalities in vital sign measurements exceeding pre-defined thresholds | Up to day 28
  Adverse event (AEs)
  Serious adverse event (SAEs)
Difference from placebo of Moxifloxacin in change from baseline (Day -1) to Day 3 at postdose extraction times for the QTcF (ΔΔQTcF) | Approximately 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Ppd Development, Llc, Austin, Texas, United States

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx